CLINICAL TRIAL: NCT05654675
Title: Evaluation of the Fractional Uptake Rate (FUR) in 18F-FDG PET/CT to Assess Tumour Metabolic Activity
Brief Title: Evaluation of the Use of the FUR to Quantify Tumor Glucose Consumption in Oncologic PET
Status: Recruiting | Type: Observational
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Roel Wierts, Medical physicist, Academisch Ziekenhuis Maastricht
Other Study IDs: NL82359.068.22
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer; Lymphoma
Keywords: PET/CT; FDG; SUV; FUR
MeSH Terms: conditions — Lung Neoplasms; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncologic patients: Lymphoma and lung cancer patients will undergo an additional dynamic FDG PET/CT examination on top of their standard care PET/CT examination.
  In addition, blood samples will be drawn at three time points
  Interventions: Diagnostic Test: FDG PET/CT

INTERVENTIONS:
Diagnostic Test: FDG PET/CT — Besides the standard care FDG PET/CT examination, subjects receive a dynamic whole body PET/CT examination.

SUMMARY:
The goal of this study is to evaluate the use of new method to quantify the amount of sugar a tumor consumes using PET/CT. The main questions it aims to answer are:

* Is the new quantification method superior with respect to the method currently used in the clinic?
* Does the new quantification method provide accurate assessment of the sugar consumption of tumours?

Participants who will undergo a standard care FDG PET/CT scan will in additional receive a dynamic PET/CT scan prior to the standard care scan. In addition blood samples will be drawn at three time points during the examination.

DETAILED DESCRIPTION:
As most tumours have a high glucose consumption, important information on tumour metabolism can be obtained from PET imaging using 18F-FDG as a radioactive glucose analogue. From literature it is known that quantitative analysis improves the clinical value of 18F-FDG PET. However, instead of measuring the true tumour glucose consumption Km, in current clinical practice the 18F-FDG uptake is measured at a certain time after administration as a surrogate for Km, the so-called standardized uptake value (SUV). As the SUV suffers from a number of important shortcomings, discrepancies between Km and the SUV have been reported which may lead to erroneous conclusions regarding disease progression based on the SUV.

Alternatively, pharmacokinetic modelling approaches facilitate accurate Km assessment. Unfortunately, these approaches typically require complex mathematical modelling, lengthy dynamic PET imaging and/or invasive arterial blood sampling and are therefore not compatible to current clinical oncologic 18F-FDG PET scanning. However, from these models it can be derived that at late time points after administration Km can be approximated using a simplified approach known as the fractional uptake rate (FUR). Our hypothesis is that the correlation between the FUR and Km is superior compared to the correlation between the SUV and Km. Therefore we expect that quantification of 18F-FDG PET images based on the FUR is superior to SUV quantifications.

The results of this study may therefore lead to a new and improved method to quantify oncologic PET images which may enhance the diagnostic value of PET. In particular, this method may lead to a more accurate assessment of tumour response to therapy and may therefore prevent continuation of unsuccessful therapy or termination of a successful therapy.

Primary objective:

To investigate whether the correlation between the FUR and Km is superior compared to the correlation between the SUV and Km.

Secondary objectives:

1. Validation of the FUR in 18F-FDG PET to accurately assess tumour metabolic activity Km.
2. To investigate the impact of the use of patient-specific versus a (scaled) population-based input function on the accuracy of Km assessment using the FUR.

The risks and patient discomfort associated with this scientific study are low. Only patients are included who already receive an 18F-FDG PET/CT scan as part of standard care.

Instead of resting on a standard hospital bed for one hour after 18F-FDG injection, patients will be resting inside the PET/CT system while a dynamic PET acquisition is performed.

In addition to their standard PET/CT examination, an extra low-dose attenuation CT scan will be performed resulting in an added radiation exposure of the patient of 3.6 mSv.

Moreover, three additional venous blood samples will be obtained at three time points, one before and two after 18F-FDG administration will be obtained from the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive an 18F FDG PET/CT scan as part of standard care
* Be competent and be 18 years of age or older

Exclusion Criteria:

* Diabetes (fasted blood glucose > 7 mmol/L)
* Not fasted > 4 hours
* Physical exercise within 24 hours
* Earlier treatment for carcinoma with radio/chemo-therapy
* Active inflammation (fever > 38 degrees, CRP > 5)
* Any condition or medical indication (such as claustrophobia) that indicates that the patient will not be able to lie still for the duration of the dynamic PET/CT examination
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 oncologic patients who will receive an 18F-FDG PET/CT scan as part of standard care will participate in this study. Therefore, recruitment of participants will take place among oncologic patients who are referred to the department of radiology and nuclear medicine of the MUMC+ for an 18F-FDG PET/CT examination.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Superiority of the FUR compared to the SUV | Time of PET examination
  The correlation between the fractional uptake rate (FUR) and the metabolic glucose consumption (Km) will be compared to the correlation between the standardized uptake value (SUV) and Km

SECONDARY OUTCOMES:
FUR validation to quantify tumour metabolic activity | Time of PET examination
  Comparison between the assessment of the tumour metabolic activity as measured by the FUR vs traditional Patlak method
Impact of patient-specific input function | Time of PET examination
  The impact of the use of a patient-specific input function is investigated compared to the use of a (scaled) population-based input function on the accuracy of Km assessment using the FUR

CONTACTS AND LOCATIONS:
Overall Officials: Roel Wierts, PhD, Principal Investigator — Medical physicist
Locations (1):
- Academisch ziekenhuis Maastricht, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided